CLINICAL TRIAL: NCT07018479
Title: Effects of a Female Hormone Balance Supplement on Premenstrual Syndrome Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VINABAS FORMULATIONS SL (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20453
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Premenstrual Syndrome
Keywords: PMS; hormonal supplement; female hormone balance
MeSH Terms: conditions — Premenstrual Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FemmeBalance Supplement Group (Experimental): Two capsules daily of FemmeBalance, containing Sabal Serrulata, NAC, turmeric extract, chasteberry extract, vitamin B5, black pepper extract, and excipients.
  Interventions: Dietary Supplement: FemmeBalance Supplement Group

INTERVENTIONS:
Dietary Supplement: FemmeBalance Supplement Group — Participants will take two capsules daily of the FemmeBalance supplement with their evening meal for four menstrual cycles

SUMMARY:
This virtual single-group study evaluates the effects of the FemmeBalance supplement on symptoms of premenstrual syndrome (PMS) over four menstrual cycles. The study involves daily intake of the supplement, regular questionnaires, and skin photo submissions for dermatological grading.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 18-40.
* Self-reported symptoms of PMS for at least three consecutive months, including but not limited to pelvic pain, mood swings, acne, hair loss, fluid retention, breast pain/tenderness, irritability, and episodes of crying or sadness.
* Generally healthy and not living with any uncontrolled chronic disease.
* Has a regular menstrual cycle between 21 and 35 days in length.
* Willing to maintain the same diet, sleep schedule, and activity level for the duration of the study (at least 16 weeks).
* Own a smartphone with a camera.
* Must reside in the United States.

Exclusion Criteria:

* Any pre-existing chronic conditions that would prevent participants from adhering to the protocol, including oncological and psychiatric disorders.
* Anyone with known severe allergic reactions that require the use of an Epi-pen or any allergies to any of the product ingredients.
* Women who are pregnant, breastfeeding, or trying to conceive.
* Anyone who is unwilling or unable to follow the study protocol.
* Anyone previously diagnosed with premenstrual dysphoric disorder (PMDD), endometriosis, or any cancer of the reproductive system.
* Anyone who is peri- or post-menopausal.
* Anyone who is currently on hormonal birth control or who has been on hormonal birth control in the last three months.
* Anyone who is taking any products, medication, or supplements that target the symptoms of PMS.
* Anyone who has undergone any surgeries or invasive treatments in the last six months or who is planning on undergoing any in the study duration.
* Anyone who has had any major illness in the last three months.
* Anyone who is currently undergoing, or who plans to undergo in the study period, any procedures relating to reproductive health and/or the menstrual cycle, e.g., a hysterectomy, ovary removal, or similar procedure.
* Anyone who suffers from amenorrhoea or irregular periods (<21 days or >35 days apart on average).
* Anyone who is currently participating in or who plans to participate in another trial during the study period.
* Anyone with a history of substance abuse.
* Anyone who smokes or who has been a smoker in the past three months.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Change in PMS Symptoms | Baseline and Day 7 of each menstrual cycle over 4 cycles (~16 weeks)
  Change in self-reported symptoms of premenstrual syndrome, including pelvic pain, mood swings, acne, hair loss, fluid retention, breast pain/tenderness, irritability, and episodes of crying or sadness, assessed using validated questionnaires (PSST and study-specific tools).

SECONDARY OUTCOMES:
Participant Perception of Supplement Effectiveness | Day 7 of each menstrual cycle over 4 cycles (~16 weeks)
  Self-reported participant feedback on perceived effectiveness of the supplement, collected through questionnaires. These responses are qualitative and not subject to statistical analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No